CLINICAL TRIAL: NCT03107221
Title: The Effectiveness and Acceptability of the Internet-based "Smart Eating" Self-help Programme Alongside Treatment as Usual for the Management of Eating Disorders: A Pilot Study
Brief Title: Eating Disorders: Online Self-help & Usual Treatment (TAU) vs TAU Only
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015MH19
Record Dates: First submitted 2016-12-12; First posted 2017-04-11 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder; Other Specified Feeding or Eating Disorder
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Access to online self-help programme "Smart Eating" along with usual treatment from a specialist eating disorder service
  Interventions: Behavioral: "Smart Eating" internet-based self-help programme
- Control (No Intervention): Usual treatment from a specialist eating disorder service

INTERVENTIONS:
Behavioral: "Smart Eating" internet-based self-help programme — An internet-based self-help programme using cognitive behavioural therapy principles to treat individuals receiving input from a specialist eating disorders service. The programme takes 3 months to complete.
  Arms: Intervention

SUMMARY:
A pilot study exploring whether individuals receiving usual treatment (CBT) from the specialist NHS Tayside Eating Disorders Service and accessing the online self-help "Smart Eating" programme have improved treatment outcomes compared to those receiving usual treatment only. The study will also explore acceptability of the "Smart Eating" self-help programme via a feedback questionnaire.

DETAILED DESCRIPTION:
This controlled-comparison pilot study will explore whether individuals receiving usual treatment (CBT) from the specialist NHS Tayside Eating Disorders Service and accessing the online self-help "Smart Eating" programme have improved treatment outcomes compared to those receiving usual treatment only. All participants would be involved in the trial for 6 months, capturing their motivation for change, eating disorder psychopathology and quality of life at four time-points (pre-treatment, mid-treatment, end of treatment, 3-month follow-up). Some participants may continue to receive usual treatment after study end, which will be detailed in the study analysis. Following trial completion, all participants will be able to access the "Smart Eating" programme. The study will also explore acceptability of the "Smart Eating" self-help programme via a feedback questionnaire to inform programme adaptations and a possible pragmatic randomised controlled trial planned for the future. Currently, no other UK study is piloting the use of the "Smart Eating" programme as an adjunct to specialist NHS eating disorder treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 16-65 years
* meet diagnostic criteria for an eating disorder
* commencing treatment under the NHS Tayside Eating Disorders Service
* fluent in English
* provide written consent
* literate to the extent of understanding self-report questionnaires & following verbal instructions
* access to a computer

Exclusion Criteria:

* deemed too emotionally or physically frail to participate by clinical staff;
* currently presenting with active suicidal intent;
* unable to read English or follow verbal English instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Improvement in eating disorder behaviours captured by the Eating Disorders Examination Questionnaire (EDE-Q) | 6 months
  Improvement will be captured by a reduction in the frequency of behaviours indicative of an eating disorder over a 28-day period across the 41-item Eating Disorders Examination Questionnaire (EDE-Q)

SECONDARY OUTCOMES:
Acceptability of "Smart Eating" programme will be captured through qualitative information gathered by a feedback questionnaire | 6 months
  Acceptability will be evaluated via a participant feedback questionnaire

OTHER OUTCOMES:
Improvement in eating psychopathology captured by the Eating Disorders Inventory 3 | 6 months
  Improvement will be captured by a reduction in symptoms indicative of an eating disorder as captured by the 91-item Eating Disorders Inventory (3 scales specific to eating disorders, 9 non-specific, general psychological scales).
Improvement in quality of life captured by an increase in scores on the SF-36 formal measure | 6 months
  Improvement in quality of life will be captured by an increase in scores on the 36-Item Short Form Health Survey (SF-36) formal measures, whereby high scores indicate good quality of life.
Change in stage of motivation for change captured by the MSCARED formal measure | 6 months
  Motivation for change is identified by the formal measure: Motivational Stage of Change for Adolescents Recovering from an Eating Disorder (MSCARED). The measure captures participants' current stage of change, and whether they play an active participation in recovery as identified by whether in the active, maintenance or recovery stage.
Reduction in symptoms of anxiety captured by the Beck Anxiety Inventory | 6 months
  Improvement will be captured by a reduction in physiological and cognitive symptoms of anxiety by the 21-item formal measure the Beck Anxiety Inventory
Reduction in symptoms of depression captured by the Beck Depression Inventory II | 6 months
  Improvement will be captured by a reduction in physiological and cognitive symptoms of depression by the 21-item formal measure the Beck Depression Inventory II.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Filgate, MSc, Principal Investigator — NHS Tayside/University of Edinburgh
Locations (1):
- NHS Tayside Eating Disorders Service, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A summary of study findings for participants are available on request